CLINICAL TRIAL: NCT00320021
Title: A Randomized, Double-Blind, Placebo-Controlled, Escalating Dose, Pilot Study to Evaluate the Safety, Tolerability and Biologic Activity of Pyridorin (Pyridoxamine Dihydrochloride) in Patients With Diabetic Nephropathy Associated With Type 1 or Type 2 Diabetes
Brief Title: Effect of Pyridorin in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioStratum (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PYR-205/207; PYR-205; PYR-207
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2006-04

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic nephropathy; Advanced Glycation Endproduct Inhibitor; Pyridorin; Pyridoxamine
MeSH Terms: conditions — Diabetic Nephropathies | interventions — pyridoxamine dihydrochloride

INTERVENTIONS:
Drug: Pyridorin (pyridoxamine dihydrochloride)

SUMMARY:
The primary objective of the study is to evaluate the safety, tolerability and efficacy of Pyridorin (pyridoxamine dihydrochloride) up to 250 mg given orally twice daily in patients with diabetic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females (non-pregnant and non-lactating) between 18 and 70 years of age with type 1 or type 2 diabetes
* Sitting blood pressure of <=170/100 mm Hg at weeks -2 and -1
* Hemoglobin A1C <=12% at week -2
* Patients with diagnosis of diabetic nephropathy as defined by

  1. Serum Creatinine <=2.0 mg/dL at weeks -2 and -1 (PYR-205) Serum Creatinine >2.0 mg/dL but <=3.5 mg/dL at weeks -2 and -1 (PYR-207)
  2. Urinary albumin excretion >=300 mg/24 hours at week -2
  3. No other known or suspected etiology for nephropathy
* Voluntary written consent to participate in this study

Exclusion Criteria:

* History of allergic or adverse response to any B vitamin
* History of major cardiovascular or cerebrovascular events
* History of cancer except adequately treated basal or squamous cell carcinoma of the skin
* History of diabetic ketoacidosis
* Autoimmune diseases
* History of significant peripheral neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2002-07; Study Completion 2003-09

PRIMARY OUTCOMES:
Change in Serum Creatinine from baseline to week 26

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten P Degenhardt, Ph.D., Study Director — BioStratum, Inc.